CLINICAL TRIAL: NCT00608140
Title: Surgery Versus Medical Treatment Alone for Patients With Significant Mitral Regurgitation and Non-ischemic Congestive Heart Failure: SMMART-HF
Brief Title: Effectiveness of Surgical Mitral Valve Repair Versus Medical Treatment for People With Significant Mitral Regurgitation and Non-ischemic Congestive Heart Failure
Acronym: SMMART-HF
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to recruit sufficient numbers of patients.
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Heart Failure Clinical Research Network (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00002860; U01HL084904 (NIH)
Record Dates: First submitted 2008-01-24; First posted 2008-02-06 (Estimated); Results first posted 2013-07-18 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2013-07

CONDITIONS: Mitral Valve Insufficiency; Heart Failure
Keywords: Advanced Heart Failure; Non-Ischemic Heart Failure; Mitral Regurgitation; Mitral Valve Replacement; Congestive Heart Failure; Surgical Mitral Valvuloplasty; Dilated Cardiomyopathy; Annular Ring
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Participants will receive optimal medical therapy plus surgical mitral valve repair with complete annular ring placement
  Interventions: Procedure: Surgical mitral valvuloplasty with placement of annular ring (SMVR); Drug: Optimal medical therapy (OMT)
- 2 (Active Comparator): Participants will receive optimal medical therapy alone
  Interventions: Drug: Optimal medical therapy (OMT)
- 3 (Experimental): Participants will receive optimal medical therapy plus 18-month delayed surgical mitral valve repair with complete annular ring placement
  Interventions: Procedure: Surgical mitral valvuloplasty with placement of annular ring (SMVR); Drug: Optimal medical therapy (OMT)

INTERVENTIONS:
Procedure: Surgical mitral valvuloplasty with placement of annular ring (SMVR) — Participants will undergo open heart surgery to mechanically reduce mitral regurgitation (MR). A complete rigid or semi-rigid annular ring will be placed unless specifically contraindicated by intraoperative findings. The ring size will be between 24 mm and 27 mm in the anteroposterior diameter. Annular ring sutures will be placed circumferentially approximately 1 mm off the hinge point between the leaflet and the atrial tissue. The total number of sutures will vary between 4 and 7 sutures anteriorly, while 8 to 12 sutures will be utilized for the posterior segment of the annulus. Additional repair of the mitral apparatus itself will be based on intraoperative findings. Leaflet repair will be performed for significant prolapse. Submitral apparatus repair will be performed for ruptured or significantly elongated chordae as well as significant chordal tethering.
  Arms: 1; 3
Drug: Optimal medical therapy (OMT) — Optimal medical therapy can include, but is not limited to, any of the following treatment regimens: combination of vasodilator therapy and diuretics, nitrates and nifedipine, and beta-adrenergic blocker therapy.

SUMMARY:
Mitral regurgitation (MR), also known as mitral insufficiency, is a condition in which the heart's mitral valve, located between two of the heart's main chambers, does not firmly shut, allowing blood to leak backwards within the heart. Improper functioning of the mitral valve disrupts the proper flow of blood through the body, resulting in shortness of breath and fatigue. When mild, MR may not pose a significant danger to a person's health, but severe MR may be associated with serious complications, such as heart failure, irregular heart rhythm, and high blood pressure. Although there are treatments for MR, including medication and surgery, more information is needed on the effectiveness of these treatments in people with significant MR. This study will compare the safety and effectiveness of corrective surgery added to optimal medical treatment (OMT) versus OMT alone in treating people with significant MR caused by an enlarged heart.

DETAILED DESCRIPTION:
It is estimated that approximately 4 out of 10 people with an enlarged heart due to heart failure develop MR, referred to as secondary MR. This type of MR is caused by enlargement of the left ventricle (LV), one of the heart's main chambers. In turn, the enlargement leads to stretching of certain heart muscles around the mitral valve and of the valve itself. Symptoms of secondary MR may include shortness of breath, fatigue, dizziness, swollen feet, cough, and heart palpitations. Mitral valve repair or replacement surgery is sometimes considered as a treatment option to restore proper heart function in people with secondary MR. Surgical repair with placement of an artificial ring around the mitral valve can help to tighten the valve and add benefit to non-surgical treatments for MR. However, although surgical placement of the ring improves mitral valve function in most people, it is not known whether this surgery helps people live longer and healthier lives. This study will compare the safety and effectiveness of surgical mitral valvuloplasty with placement of an annular ring (SMVR) added to optimal medical treatment (OMT) versus OMT alone in non-ischemic heart failure patients with significant secondary MR.

Participation from baseline through follow-up in this study will last 18 months. All potential participants will initially undergo a transesophageal echocardiogram to confirm the presence of an abnormal mitral valve. Eligible participants will then undergo a number of baseline tests, which will include cardiopulmonary exercise stress testing, a chest wall echocardiogram, blood draw, 6-minute walk test, medical questionnaires, and a physical exam. Next, participants will be randomly assigned to receive immediate open heart surgery with the placement of a mitral valve ring, delayed surgery at least 18 months later, or OMT. Participants assigned to receive immediate surgery will undergo the surgery 2 weeks after baseline testing. Participants assigned to receive OMT will receive treatment with any of the following medication regimens: combination of vasodilator therapy and diuretics, nitrates and nifedipine, and beta-adrenergic blocker therapy. Follow-up visits for all participants will occur at Months 1, 3, 6, 12, and 18 and will include repeat baseline testing. Long-term survival status data may be collected beyond 18 months for some participants.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic chronic heart failure, New York Heart Association (NYHA) class II to IIIb
* Left ventricular ejection fraction of 0.35 due to non-ischemic etiology
* Evidence by transthoracic echocardiography (TTE) of moderate or severe MR without obvious primary mitral valve pathology
* Peak VO2 less than or equal to 22 ml/kg/min, as obtained at study entry
* Optimal heart failure therapy for at least 6 months prior to study entry

Exclusion Criteria:

* Significant coronary artery disease (greater than 75% lesion in any vessel) by coronary angiography or by a history of a prior heart attack
* Heart failure due to active myocarditis, congenital heart disease, or obstructive hypertrophic cardiomyopathy
* Significant ventricular arrhythmias not treated with an implantable defibrillator
* Primary MR due to significant chordal or leaflet abnormalities by TTE
* Other hemodynamically relevant stenotic or regurgitant valvular diseases
* Severe tricuspid regurgitation (TR) (moderate TR is allowed)
* Severe pulmonic regurgitation (PR) (moderate PR is allowed)
* Moderate to severe aortic regurgitation
* Any moderate to severe stenotic lesions using American Heart Association/American College of Cardiology (AHA/ACC) criteria 31
* Dependence on chronic inotropic therapy
* Restrictive cardiomyopathy or constrictive pericarditis
* Severe right ventricular dysfunction
* Baseline creatinine greater than or equal to 3 mg/dL or renal replacement therapy (chronic hemodialysis or peritoneal dialysis)
* Poor transthoracic sonographic windows precluding reasonable assessment of LV endocardial borders from apical imaging on TTE
* Inability to perform the spirometric exercise testing
* Significant chronic lung disease that might interfere with the ability to interpret the spirometric measurements, including home oxygen, forced expiratory volume in 1 second (FEV1) less than 1.0 L/min, or exertional hypoxemia with saturations less than 90%
* Any known neoplastic disease other than skin cancer
* Other terminal illness with a life expectancy less than 1 year
* Plan for percutaneous mitral valve procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry L. Lee, PhD, Principal Investigator — Duke Clinical Research Institute; Eugene Braunwald, MD, Study Chair — Harvard University
Locations (9):
- United States (8):
  - Morehouse School of Medicine, Atlanta, Georgia
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Minnesota Heart Failure Network, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - Baylor College of Medicine, Houston, Texas
  - University of Utah Health Sciences Center, Murray, Utah
  - University of Vermont - Fletcher Allen Health Care, Burlington, Vermont
- Montreal Heart Institute, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- 1 Medical Therapy Plus Surgery: Participants will receive optimal medical therapy plus surgical mitral valve repair with complete annular ring placement
- 2 Medical Therapy Only: Participants will receive optimal medical therapy alone
Period: Overall Study
Arm/Group | 1 Medical Therapy Plus Surgery | 2 Medical Therapy Only
Started | 1 | 1
Completed | 0 (Study ended early due to low enrollment) | 0 (Study ended early due to low enrollment)
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- 1 Medical Therapy Plus Surgical Repair: Participants will receive optimal medical therapy plus surgical mitral valve repair with complete annular ring placement
- Total: Total of all reporting groups
Arm/Group | 1 Medical Therapy Plus Surgical Repair | 2 Medical Therapy Only | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — Standard deviation for individual arms could not be calculated because only 1 participant was evaluated in each arm. Total SD was calculated.
  years | 65.5 | 63 | 64.25 (1.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Effect of Adding SMVR to OMT Alone on LV Remodeling, Specifically LV End-systolic Volume Index (LVESVI)
Time Frame: Measured at Month 18
Population: Data were not analyzed due to study termination
Arm/Group | 1 Medical Therapy Plus Surgery | 2 Medical Therapy Only
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Peak VO2
Time Frame: Measured at Month 18
Population: The 2 patients enrolled in the study did not reach their endpoints before the trial was closed. No data were collected for this outcome measure and no analysis was performed.
Groups:
- Optimal Medical Therapy Plus Surgical MV Repair: Participants will receive optimal medical therapy plus surgical mitral valve repair with complete annular ring placement
  Surgical mitral valvuloplasty with placement of annular ring (SMVR): Participants will undergo open heart surgery to mechanically reduce mitral regurgitation (MR). A complete rigid or semi-rigid annular ring will be placed unless specifically contraindicated by intraoperative findings. Additional repair of the mitral apparatus itself will be based on intraoperative findings. Leaflet repair will be performed for significant prolapse. Submitral apparatus repair will be performed for ruptured or significantly elongated chordae as well as significant chordal tethering.
- Optimal Medical Therapy Alone: Participants will receive optimal medical therapy alone
  Optimal medical therapy (OMT): Optimal medical therapy can include, but is not limited to, any of the following treatment regimens: combination of vasodilator therapy and diuretics, nitrates and nifedipine, and beta-adrenergic blocker therapy.
- Optimal Medical Therapy Plus 18 Month Delayed MVR: Participants will receive optimal medical therapy plus 18-month delayed surgical mitral valve repair with complete annular ring placement
  Surgical mitral valvuloplasty with placement of annular ring (SMVR): Participants will undergo open heart surgery to mechanically reduce mitral regurgitation (MR). Additional repair of the mitral apparatus itself will be based on intraoperative findings. Leaflet repair will be performed for significant prolapse. Submitral apparatus repair will be performed for ruptured or significantly elongated chordae as well as significant chordal tethering.
Arm/Group | Optimal Medical Therapy Plus Surgical MV Repair | Optimal Medical Therapy Alone | Optimal Medical Therapy Plus 18 Month Delayed MVR
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change in 6-minute Walk Test
Description: The 2 patients enrolled did not meet the 18 month measurement of primary/secondary endpoints before the trial was terminated. No data were collected for this outcome measure and no analysis was performed.
Time Frame: Measured at baseline and Month 18 but n/a
Population: The 2 patients enrolled did not meet the 18 month measurement of primary/secondary endpoints before the trial was terminated. No data were collected for this outcome measure and no analysis was performed.
Groups:
- Optimal Medical Therapy Plus Surgical MVR: Participants will receive optimal medical therapy plus surgical mitral valve repair with complete annular ring placement
  Surgical mitral valvuloplasty with placement of annular ring (SMVR): Participants will undergo open heart surgery to mechanically reduce mitral regurgitation (MR). Additional repair of the mitral apparatus itself will be based on intraoperative findings. Leaflet repair will be performed for significant prolapse. Submitral apparatus repair will be performed for ruptured or signific
- Optimal Medical Therapy Plus 18 Month Delayed MVR: Participants will receive optimal medical therapy plus 18-month delayed surgical mitral valve repair with complete annular ring placement
  Surgical mitral valvuloplasty with placement of annular ring (SMVR): Participants will undergo open heart surgery to mechanically reduce mitral regurgitation (MR). Additional repair of the mitral apparatus itself will be based on intraoperative findings. Leaflet repair will be performed for significant prolapse. Submitral apparatus repair will be performed for rup
Arm/Group | Optimal Medical Therapy Plus Surgical MVR | Optimal Medical Therapy Alone | Optimal Medical Therapy Plus 18 Month Delayed MVR
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change in Minnesota Living With Heart Failure (MLHF) Score
Description: Change in MLHF score. However, the 2 patients enrolled did not meet the 18 month measurement of primary/secondary endpoints before the trial was terminated. No analysis was performed.
Time Frame: Planned to be measured at baseline and Month 18 but n/a
Population: as for outcome 3
Groups:
- Optimal Medical Therapy Plus Surgical MVR: Participants will receive optimal medical therapy plus surgical mitral valve repair with complete annular ring placement
  Surgical mitral valvuloplasty with placement of annular ring (SMVR): Participants will undergo open heart surgery to mechanically reduce mitral regurgitation (MR). Additional repair of the mitral apparatus itself will be based on intraoperative findings. Leaflet repair will be performed for significant prolapse. Submitral apparatus repair will be performed for ruptured or significantly elongated chordae as well as significant chordal tethering.
  Optimal medical therapy (OMT): Optimal medical therapy can include, but is not limited to, any of the following treatment regimens: combination of vasodilator therapy and diuretics, nitrates and nifedipine, and beta-adrenergic blocker therapy.
- Optimal Medical Therapy Plus 18 Month Delayed MVR: Participants will receive optimal medical therapy plus 18-month delayed surgical mitral valve repair with complete annular ring placement
  Surgical mitral valvuloplasty with placement of annular ring (SMVR): Participants will undergo open heart surgery to mechanically reduce mitral regurgitation (MR). Additional repair of the mitral apparatus itself will be based on intraoperative findings. Leaflet repair will be performed for significant prolapse. Submitral apparatus repair will be performed for ruptured or significantly elongated chordae as well as significant chordal tethering.
  Optimal medical therapy (OMT): Optimal medical therapy can include, but is not limited to, any of the following treatment regimens: combination of vasodilator therapy and diuretics, nitrates and nifedipine, and beta-adrenergic blocker therapy.
Arm/Group | Optimal Medical Therapy Plus Surgical MVR | Optimal Medical Therapy Alone | Optimal Medical Therapy Plus 18 Month Delayed MVR
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Total Days Alive and Total Days Not Hospitalized
Description: Total days alive and not hospitalized by 18 months. However, the 2 patients enrolled did not meet the 18 month measurement of primary/secondary endpoints before the trial was terminated. No analysis was performed.
Time Frame: Measured at baseline and Month 18
Population: as for outcome 3
Arm/Group | Optimal Medical Therapy Plus Surgical MVR | Optimal Medical Therapy Alone | Optimal Medical Therapy Plus 18 Month Delayed MVR
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Total Mortality (All Causes)
Description: Total all-cause mortality at 18 months. However, the 2 patients enrolled did not meet the 18 month measurement of primary/secondary endpoints before the trial was terminated. No analysis was performed.
Time Frame: Measured at Month 18
Population: as for outcome 3
Groups:
- Optimal Medical Therapy Plus Surgical MVR: Participants will receive optimal medical therapy plus surgical mitral valve repair with complete annular ring placement
  Surgical mitral valvuloplasty with placement of annular ring (SMVR): Participants will undergo open heart surgery to mechanically reduce mitral regurgitation (MR). A complete rigid or semi-rigid annular ring will be placed unless specifically contraindicated by intraoperative findings. Additional repair of the mitral apparatus itself will be based on intraoperative findings. Leaflet repair will be performed for significant prolapse. Submitral apparatus repair will be performed for ruptured or significantly elongated chordae as well as significant chordal tethering.
  Optimal medical therapy (OMT): Optimal medical therapy can include, but is not limited to, any of the following treatment regimens: combination of vasodilator therapy and diuretics, nitrates and nifedipine, and beta-adrenergic blocker therapy.
- Optimal Medical Therapy Plus 18 Month Delayed MVR: Participants will receive optimal medical therapy plus 18-month delayed surgical mitral valve repair with complete annular ring placement
  Surgical mitral valvuloplasty with placement of annular ring (SMVR): Participants will undergo open heart surgery to mechanically reduce mitral regurgitation (MR). A complete rigid or semi-rigid annular ring will be placed unless specifically contraindicated by intraoperative findings. Additional repair of the mitral apparatus itself will be based on intraoperative findings. Leaflet repair will be performed for significant prolapse. Submitral apparatus repair will be performed for ruptured or significantly elongated chordae as well as significant chordal tethering.
  Optimal medical therapy (OMT): Optimal medical therapy can include, but is not limited to, any of the following treatment regimens: combination of vasodilator therapy and diuretics, nitrates and nifedipine, and beta-adrenergic blocker therapy.
Arm/Group | Optimal Medical Therapy Plus Surgical MVR | Optimal Medical Therapy Alone | Optimal Medical Therapy Plus 18 Month Delayed MVR
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Perioperative Mortality
Time Frame: Measured between Days 0 and 30 postsurgery
Measure: Number; unit: participants
Arm/Group | 1 Medical Therapy Plus Surgery | 2 Medical Therapy Only
Number analyzed (Participants) | 1 | 1
participants | 0 | 0

ADVERSE EVENTS:
Description: Adverse events were not collected, only serious adverse events were collected. "0" was entered for Total Number of Participants at Risk where Adverse events were not collected.
Arm/Group | 1 Medical Therapy Plus Surgery | 2 Medical Therapy Only
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Medical Therapy Plus Surgery (N=1) | 2 Medical Therapy Only (N=1)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 1 (1)
HAEMODYNAMIC INSTABILITY (Cardiac disorders) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No